CLINICAL TRIAL: NCT05418738
Title: The Relationship Between Psychosocial Factors Affecting Pain Perception and Physical Activity Level in Pregnant Women With Lumbopelvic Pain
Status: Completed | Type: Observational
Sponsor: Uskudar University (Other)
Responsible Party: Principal Investigator, tuba kolaylı, Lecturer, Uskudar University
Other Study IDs: Uskudar University
Record Dates: First submitted 2022-06-09; First posted 2022-06-14 (Actual); Last update posted 2022-06-14 (Actual); Status verified 2022-06

CONDITIONS: Investigate the Relationship Between the Psychosocial Factors Affecting Pain Perception and Physical Activity Levels in Pregnant Women With Lumbopelvic Pain
Keywords: lumbopelvic pain, psychosocial features, physical activity, pelvic pain, pregnancy
MeSH Terms: conditions — Motor Activity; Pelvic Pain

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Lumbopelvic pain (LPP) is a common condition encountered during pregnancy. During pregnancy, 50% of women experience LPP. This study was planned to show the relationship between psychosocial factors affecting the perception of pain such as pregnancy-related psychosocial factors, pregnancy-related distress, catastrophization and pain self-efficacy and physical activity level in pregnant women with lumbopelvic pain. This study was conducted using the questionnaires.

DETAILED DESCRIPTION:
In pregnant women with lumbopelvic pain, physical activity during pregnancy has many positive effects on both maternal and infant health. Therefore, it is necessary to know the factors affecting physical activity during pregnancy and make arrangements regarding these factors. This study was planned to reveal the relationship between pregnancy-related psychosocial factors, pregnancy-related distress, catastrophizing, and pain self-efficacy, which affect pain perception, and physical activity level in pregnant women with lumbopelvic pain. The study was conducted with 60 pregnant women who met the inclusion criteria. This study was conducted using the questionnaires prepared in the electronic environment and sent to the participants. This study aims to investigate the relationship between the psychosocial factors affecting pain perception and physical activity levels in pregnant women with LPP.

ELIGIBILITY:
Inclusion Criteria:

* Women between the ages of 18-45, who had pain in the lumbopelvic region for more than a week, who had pain between 1-10 according to the VAS, who could read and understand Turkish, who were in the second or third trimester of pregnancy, and who did not exercise regularly before pregnancy were included in this cross-sectional and descriptive study.

Exclusion Criteria:

* having pregnancy complications (preeclampsia, pregnancy-related hypertension, diabetes, etc.), having gynecological or urological problems leading to pain during pregnancy, and having a history of acute or chronic disease, surgical intervention and trauma in the musculoskeletal or nervous system.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Pregnant women between the ages of 18-45, who had lumbopelvic pain
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
The Antenatal Psychosocial Health Assessment Scale (ALPHA) | 20 munites
  ALPHA was used to evaluate the psychosocial states of pregnant women participating in the study. The ALPHA was created by Yıldız in 2011 to assess the psychosocial health states of pregnant women.
Tilburg Pregnancy Distress Scale (TPDS) | 10 minutes
  TPDS, was used to determine the distress states of pregnant women. The TPDS is used to assess distress developing during pregnancy. The TPDS, which was created by Pop et al. in 2011, consists of 16 items in total.
Pain Catastrophizing Scale (PCS) | 10 munites
  PCS, was used to determine ehe level of pain catastrophizing in pregnant women. It was developed by Sullivan et al. in 1995 to assess the exaggerated and negative mental response of individuals during the pain experience, in other words, their levels of catastrophizing. The PCS is comprised of 13 items, including the feelings and opinions of individuals about their last pain experience.
The Pain Self-Efficacy Questionnaire (PSEQ) | 5 munites
  PSEQ applied to the participating pregnant women was created by M.K. Nicholas in 1989 to assess the confidence of individuals, who experienced pain, in carrying out activities despite pain. It consists of 10 items.
The Pregnancy Physical Activity Questionnaire (PPAQ) | 20 minutes
  PPAQ was used to reveal the physical activity levels of pregnant women. With this questionnaire, the intensity, frequency, and duration of physical activity are evaluated in pregnant women. It consists of 32 items that assess housework/caregiving activities, professional activities, sports/exercise activities, transportation activities, and inactivity.

CONTACTS AND LOCATIONS:
Locations (1):
- Uskudar University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided